CLINICAL TRIAL: NCT07382466
Title: Workstation Ergonomics Intervention to Reduce Musculoskeletal Symptoms Among University Employees
Brief Title: Workstation Ergonomics Program at Al-Baha University
Acronym: ERG-ABU
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Baha University (Other)
Responsible Party: Principal Investigator, Dr. Wael Alghamdi, Associate Professor، Dean, College of Nursing، Consultant Physiotherapist, Al-Baha University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 46120176/2025
Record Dates: First submitted 2026-01-27; First posted 2026-02-02 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Work-Related Musculoskeletal Disorders; Musculoskeletal Disorders; Occupational Musculoskeletal Disorders
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Intervention Model Description: Two-arm parallel-group study (intervention vs control) with pre-post assessments.
Masking Description: Open-label; no masking was implemented.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ergonomics Program (Intervention) (Experimental): Participants will receive an office-workstation ergonomics program including a self-assessment checklist-based evaluation and tailored recommendations for workstation adjustment and safe working posture, along with brief educational guidance and periodic follow-up reminders during the study period.
  Interventions: Behavioral: Workstation Ergonomics Program
- Usual Practice (Control) (Active Comparator): Participants will continue their usual workstation practices during the study period and will not receive the ergonomics recommendations/education until after completion of follow-up assessment.
  Interventions: Behavioral: Usual Practice (Control)

INTERVENTIONS:
Behavioral: Workstation Ergonomics Program — Participants in the intervention arm will complete an online computer workstation self-assessment checklist. Based on their responses, they will receive individualized workstation ergonomics guidance and educational materials covering optimal sitting posture and workstation setup (chair/desk height, monitor position, keyboard/mouse placement, and lighting), as well as recommendations for regular micro-breaks and simple stretching. Guidance will be delivered electronically after baseline assessment, and participants will be encouraged to implement the recommendations throughout the follow-up period (4 weeks) with reinforcement reminders.
  Other Names: Ergonomics Education and Workstation Self-Assessment
  Arms: Ergonomics Program (Intervention)
Behavioral: Usual Practice (Control) — Participants in the control arm will receive no ergonomics training, individualized recommendations, or educational materials during the study period and will continue their usual computer workstation practices. After completion of follow-up assessments, the control group will be offered the same ergonomics educational materials and general workstation guidance provided to the intervention arm.
  Arms: Usual Practice (Control)

SUMMARY:
This study evaluates a workstation ergonomics program at Al-Baha University aimed at reducing work-related musculoskeletal symptoms among university employees who use computers regularly. The program includes an ergonomics self-assessment of the workstation, individualized guidance on proper workstation setup and posture, and practical recommendations to improve daily work habits. Participants will be followed for approximately four weeks, and changes in musculoskeletal symptoms and related outcomes will be assessed before and after the program, compared with a usual-practice control group.

DETAILED DESCRIPTION:
This is a controlled, non-randomized pre-post study conducted among university employees at Al-Baha University. Eligible participants will be allocated to either an ergonomics intervention group or a usual-practice control group. The intervention consists of a structured workstation ergonomics package that includes: (1) completing a validated workstation self-assessment checklist, (2) receiving individualized feedback and practical recommendations to optimize workstation arrangement and working posture, and (3) brief reminders to support adherence during the follow-up period. Assessments will be performed at baseline and at the end of follow-up (approximately four weeks). The primary objective is to determine whether the ergonomics program is associated with improvement in musculoskeletal symptoms compared with the control condition under real-world workplace settings.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-55 years.
* Affiliated with Al-Baha University (staff, or faculty) and regularly use a computer workstation (≥3 hours/day or ≥15 hours/week).
* Able to read and complete the online questionnaire and provide informed consent.

Exclusion Criteria:

* Current severe musculoskeletal disorder or recent major injury/surgery that markedly limits daily activities or requires ongoing medical treatment.
* Diagnosed neurological or rheumatologic condition affecting the musculoskeletal system (e.g., severe radiculopathy, inflammatory arthritis).
* Pregnancy (if you prefer to exclude it).
* Participation in another ergonomics intervention program during the study period.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-02-10 (Estimated); Primary Completion 2026-02-10 (Estimated); Study Completion 2026-04-10 (Estimated)

PRIMARY OUTCOMES:
Change in musculoskeletal symptoms (Nordic Musculoskeletal Questionnaire [NMQ]) | Baseline and 4 weeks.
  Change from baseline in musculoskeletal symptom burden measured using the Nordic Musculoskeletal Questionnaire (NMQ). The outcome will be calculated as the number of body regions with self-reported musculoskeletal symptoms (Yes/No) during the last 12 months, summed across assessed regions (range: 0 to 8, where 0 = no symptoms in any region and 8 = symptoms in all regions). Higher values indicate worse musculoskeletal symptoms. Outcomes will be compared between the intervention and control arms.

SECONDARY OUTCOMES:
Change in workstation ergonomics score (Computer Workstation Ergonomics: Self-Assessment Checklist) | Baseline and 4 weeks
  Change from baseline in workstation ergonomics measured using the Computer Workstation Ergonomics: Self-Assessment Checklist. The outcome will be calculated as the total checklist score, summed across all items (range: 0 to 20), where higher scores indicate better workstation ergonomics (better setup). Outcomes will be compared between the intervention and control arms.

IPD SHARING:
Plan to Share IPD: No